CLINICAL TRIAL: NCT05044039
Title: Phase I Dose Escalation and Dose Expansion Study of Duvelisib Following Chimeric Antigen Receptor T-Cell Therapy
Brief Title: Duvelisib Following Chimeric Antigen Receptor T-Cell Therapy
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: SecuraBio (Industry); The Foundation for Barnes-Jewish Hospital (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 202111018; 5R35CA210084 (NIH)
Record Dates: First submitted 2021-09-03; First posted 2021-09-14 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Non-hodgkin Lymphoma; Acute Lymphocytic Leukemia
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — duvelisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dose Escalation Stage: Duvelisib (Experimental): * Duvelisib is an oral medication taken on a once or twice daily basis on all dosing days. Doses being explored in this study are 15 mg BID (starting dose), 25 mg BID, and 15 mg QD. In the dose escalation stage, patients will receive duvelisib from Day -2 through Day 28.
  * CAR T-cells will be given per standard of care.
  Interventions: Drug: Duvelisib
- Cohort A Dose Expansion Stage: Duvelisib (Experimental): * Patients in Cohort A will receive duvelisib from Day -2 to Day 28. The dose that will be given will be determined in the dose escalation stage (the maximum tolerated dose).
  * CAR T-cells will be given per standard of care.
  Interventions: Drug: Duvelisib
- Cohort B Dose Expansion Stage: Duvelisib (Experimental): * Patients in Cohort B will receive duvelisib from Day -2 to Day 180 as follows:
    * Cycle 1 dosing begins on Day -2 and continues through Day 28 followed by 2 weeks off therapy
    * Cycles 2-6 are 28 days long and consist of dosing on Days 1 through 14, with 2 weeks off therapy.
  * CAR T-cells will be given per standard of care.
  Interventions: Drug: Duvelisib

INTERVENTIONS:
Drug: Duvelisib — Patients should take duvelisib at approximately the same time every day, with or without food.

SUMMARY:
While chimeric antigen receptor T-cell (CAR T-cell) therapy produces impressive response rates in heavily pre-treated patients, early loss of response remains a barrier. One potential mechanism of relapse is limited CAR T-cell persistence. Pre-clinical research shows that PI3K inhibition represents an intriguing mechanism for increasing CAR T-cell persistence that is easily reversible and CAR T-cell agnostic. The investigators hypothesize that PI3K inhibition with duvelisib would be safe, may provide effective prophylaxis against cytokine release syndrome (CRS), and may enhance the persistence and efficacy of CAR T-cells in the treatment of hematologic malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Meets FDA-approved criteria for treatment of non-Hodgkin lymphoma (NHL) with axicabtagene ciloleucel (Yescarta), tisagenlecleucel (Kymriah), lisocabtagene maraleucel (Breyanzi) or brexucabtagene autoleucel (Tecartus). Subjects receiving breuxacabtagene autoleucel for treatment of B-cell acute lymphoblastic leukemia (ALL) are not eligible.
* At least 18 years of age.
* The effects of duvelisib on the developing human fetus are unknown. For this reason, women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry, for the duration of study participation, and for at least 3 months after the last dose of duvelisib, as well as conform to institutional CAR T-cell guidelines. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of the study, and for at least 3 months after the last dose of duvelisib.
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

* Receiving axicabtagene ciloleucel, tisagenlecleucel, lisocabtagene maraleucel, or brexucabtagene autoleucel for the treatment of B-cell acute lymphoblastic leukemia.
* Known allergy or intolerance to duvelisib or another PI3K inhibitor. Previous treatment with duvelisib or other PI3K inhibitor is permitted unless therapy was discontinued due to toxicity or intolerance of therapy.
* Receiving therapy with a strong CYP3A inducer or inhibitor that cannot be discontinued during duvelisib therapy. Subjects receiving a strong CYP3A inducer or inhibitor at screening are eligible to participate if the drug can be discontinued the longest of the following time periods prior to initiation of duvelisib: 7 days (for strong CYP3A inhibitors), 14 days (for strong CYP3A inducers) or 4-5 half-lives (either inducer or inhibitor).
* Active CNS involvement by hematologic malignancy under treatment
* Evidence of uncontrolled infection of any origin (viral, bacterial, or fungal)
* Active bacterial, fungal or mycobacterial infection tuberculosis requiring treatment within the two years prior to study enrollment
* Known HIV infection, untreated hepatitis C or hepatitis B infection. Untreated hepatitis B is not an exclusion if hepatitis B is undetectable.
* Acute or chronic GVHD requiring systemic therapy
* Concurrent use of chronic systemic steroids or immunosuppressant medications
* Known history of immunologic/autoimmune disease affecting the CNS unrelated to diagnosis of hematologic malignancy under treatment
* Clinically significant pulmonary disease, defined as grade 2 or greater dyspnea or grade 2 or greater hypoxia
* Clinically significant cardiac disease, defined as unstable angina, acute myocardial infarction in the last 6 months, and NYHA class II or IV heart failure. Subjects with unstable arrhythmias that are not stable with medical management in 2 weeks prior to day -2 are also excluded.
* Clinically significant hepatic disease, defined as ALT, AST or alkaline phosphatase ≥ 3x ULN or total bilirubin > 1.5x ULN (unless related to Gilbert's or Meulengracht's syndrome). Subjects with a history of chronic liver disease, previous veno-occlusive disease, active alcohol abuse or history of alcohol abuse within the past 6 months are also excluded.
* Clinically significant renal disease, defined as calculated or measured creatinine clearance < 50 mL/min
* Currently breastfeeding or pregnant. Women of childbearing potential must have a negative pregnancy test within 7 days of study entry.
* Inability to swallow and retain oral medication or prior surgery or GI dysfunction that may affect drug absorption (i.e. gastric bypass surgery, gastrectomy)
* Receipt of a prior investigational agent within 4 weeks before Day -3 or currently receiving any other investigational agents.
* Unable to receive prophylactic treatment for pneumocystis, HSV or VZV at screening
* Any condition that would, in the investigator's judgment, interfere with full participation in the study, including administration of medication, attendance of study visits, elevated risk of complications or interference with interpretation of the study data
* A history of other malignancy with the exception of malignancies for which all treatment was completed at least 2 years before registration and the patient has no evidence of disease. Non-metastatic, non-melanoma skin cancers are not considered exclusionary.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2022-02-28 (Actual); Primary Completion 2026-01-06 (Actual); Study Completion 2030-05-22 (Estimated)

PRIMARY OUTCOMES:
Toxicity as measured by number of adverse events | From start of treatment through 30 days after completion of duvelisib (up to day 60 for Cohort A and up to day 212 for Cohort B)
  Toxicity is graded using NCI CTCAE v 5.0

SECONDARY OUTCOMES:
Cumulative incidence of cytokine release syndrome (CRS) | By Day 28
  -Any and grade 3-4 per ASTCT criteria
Cumulative incidence of immune effector cell-associated neurotoxicity syndrome (ICANS) | By Day 28
  -Any and grade 3-4 per ASCT criteria
Number of participants who receive anti-IL-6 agents for treatment of cytokine release syndrome (CRS) | Through completion of follow-up (estimated to be 6 months)
Number of participants who receive steroids for treatment of cytokine release syndrome (CRS) | Through completion of follow-up (estimated to be 6 months)
Number of participants with complete response (CR) | At 1 month
Number of participants with complete response (CR) | At 3 months
Number of participants with complete response (CR) | At 6 months
Best overall response rate | At 1 month
  -Defined as proportion of subjects with complete response (CR) or partial response (PR) by Lugano criteria
Best overall response rate | At 3 months
  -Defined as proportion of subjects with complete response (CR) or partial response (PR) by Lugano criteria
Best overall response rate | At 6 months
  -Defined as proportion of subjects with complete response (CR) or partial response (PR) by Lugano criteria
Progression-free survival (PFS) | Through completion of follow-up (estimated to be 5 years)
Overall survival (OS) | Through completion of follow-up (estimated to be 5 years)
Proportion of participants with partial response (PR) on Day 30 with improved response on Day 90 | Day 90
Proportion of participants with partial response (PR) on Day 30 with improved response on Day 180 | Day 180

CONTACTS AND LOCATIONS:
Overall Officials: Armin Ghobadi, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

DOCUMENTS (1):
  • Informed Consent Form (2025-06-11): https://cdn.clinicaltrials.gov/large-docs/39/NCT05044039/ICF_000.pdf